CLINICAL TRIAL: NCT05064722
Title: Initial Safety and Device Functionality of the Self-Forming Magnetic Anastomosis Device to Create a Duodenal-Ileal Diversion in Obese Patients Undergoing Primary Sleeve (SNAP-S) or Those With Inadequate Weight Loss After Sleeve (SNAP-PS)
Brief Title: Duodenal-Ileal Diversion in Obese Patients Undergoing Primary Sleeve or Those With Inadequate Weight Loss After Sleeve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GI Windows, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIW 21-001
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-06

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- SNAP-S (Experimental): Creation of a D-I diversion in participants undergoing primary sleeve gastrectomy (SNAP-S cohort)
  Interventions: Device: Self Forming Magnets (SFM)
- SNAP-PS (Experimental): Creation of a D-I diversion in participants who have experienced inadequate weight loss following sleeve gastrectomy (SNAP-PS cohort)
  Interventions: Device: Self Forming Magnets (SFM)

INTERVENTIONS:
Device: Self Forming Magnets (SFM) — To create the duodenal-ileal diversion, the duodenal magnet will be placed transorally in the proximal duodenum and the distal magnet will be placed in the ileum. Magnets are coupled and a compression induced anastomosis is created.

SUMMARY:
The objectives of this study are to assess the initial safety and device functionality of the SFM Anastomosis System including delivery systems when used to create a dual-path duodenal-ileal (D-I) diversion either during sleeve gastrectomy (i.e., SNAP-S procedure) or patients with prior sleeve gastrectomy who experience inadequate weight loss (i.e., SNAP-PS procedure). Additionally, the study is designed to evaluate the potential of the SNAP-S/SNAP-PS procedures to induce weight loss and to improve metabolic comorbidities in obese subjects.

DETAILED DESCRIPTION:
This is a single-arm, single-center, early feasibility study to evaluate the use of the SFM Anastomosis System for creation of a D-I diversion in participants undergoing primary sleeve gastrectomy (SNAP-S cohort) or who have experienced inadequate weight loss following sleeve gastrectomy (SNAP-PS cohort) defined to be failure to achieve a minimum 50% EWL at least 18 months post sleeve gastrectomy. Five patients will be enrolled in each cohort. Adult male and female subjects between the ages of 22 and 65 years-old who are candidates for the primary or revisional surgery will be considered for participation.

Patients appearing to meet basic eligibility criteria and who sign the study specific consent form will be screened for enrollment into this study and will be assessed by a multidisciplinary research team with pre-procedure nutritional and medical evaluation (including psychological and behavioral evaluation by an internist/bariatrician).

Subjects meeting the inclusion and exclusion criteria and enrolled into the study will undergo a dual-path enteral diversion using the SFM anastomosis device in which the duodenum will be connected to the ileum with the creation of a side-by-side anastomosis using the SFM device and delivery systems. For subjects undergoing concurrent sleeve gastrectomy and D-I Diversion (SNAP-S cohort) it is anticipated that the D-I diversion will be created first followed by the sleeve gastrectomy (unless the investigator determines that the reverse order is more appropriate for a particular subject).

ELIGIBILITY:
Inclusion Criteria:

1. Age 22-65 years at screening
2. Obesity with Body Mass Index (BMI) ≥ 35 kg/m2 with at least one obesity related comorbidity or ≥ 40 but ≤ 50 kg/m2 with or without comorbidities at time of screening.

   a. For SNAP-PS Cohort, subject should be at least 18 months from the initial sleeve gastrectomy and have failed to achieve at minimum 50% EWL
3. If subject has obesity-related comorbidities such as hypertension, dyslipidemia, and sleep apnea, these comorbidities must be well-controlled.
4. Able to understand and sign informed consent document
5. Patient lives, and intends to remain, within a 300-km radius of study center for 24 months
6. Willing to refrain from smoking during the study follow-up period
7. If subject is female, she must commit to not becoming pregnant for 24 months and agree to use of contraceptives during this period and may not be nursing

Exclusion Criteria:

1. Type 1 Diabetes
2. Uncontrolled T2DM Fasting glucose ≥ 200 mg/dl (11.1 mmol/L) and/or hemoglobin A1c >10 or use of injectable insulin
3. Any documented conditions for which endoscopy and/or laparoscopy would be contraindicated or history of previous technically difficult or failed endoscopy
4. Contraindication to general anesthesia
5. Clinically significant finding during procedural endoscopy such as presence of an unhealed ulcers, bleeding lesions, tumors or ischemic or necrotic tissue at target magnet deployment site
6. Congenital or acquired anomalies of the GI tract, including atresias, stenosis, prior obstruction or malrotation
7. Presence of a duodenal diverticulum (>10mm)
8. Any previous major surgery on the stomach, duodenum, hepatobiliary tree (excluding laparoscopically removed gallbladder or prior sleeve gastrectomy for SNAP-PS cohort), pancreas or right colon
9. History of chronic gastrointestinal disease (e.g., cirrhosis, inflammatory bowel disease) that in the opinion of the Investigator may preclude safe and complete study participation
10. Uncontrolled severe hypertension (blood pressure >160/100mmHg)
11. Pre-existing severe comorbid cardio-respiratory disease (e.g., congestive heart failure, uncontrolled cardiac arrhythmia, coronary artery disease, chronic obstructive lung disease requiring supplemental oxygen, pulmonary embolism, MI with prior 6 months)
12. Liver biochemistries (ALT and AST) ≥ 3 times the upper limit of normal
13. Uncorrectable coagulation disorder (platelets < 100,000, PT >2 seconds above control or INR >1.5) at time of procedure, Note: management of anti-platelet medications, when applicable, will follow standard practices of the institution
14. Uncorrectable anemia (Hemoglobin < 11 g/dL in women and <12.5 g/dL in men)
15. Specific genetic or hormonal cause of obesity such as Prader -Willi syndrome
16. For females of child-bearing potential: Pregnancy or desire to be pregnant during the study

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-10-09 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 12 months
  Total Body Weight Loss from baseline

SECONDARY OUTCOMES:
Percent Responders | 12 Months
  Percent of patients losing at least 10% of their baseline weight
%EWL | 12 Months
  Mean Excess Weight Loss from baseline
Serum lipids | 12 Months
  Mean change of serum lipids from baseline
Systolic/diastolic blood pressure | 12 Months
  Mean percent change in systolic/diastolic blood pressure from baseline
Hemoglobin A1c | 12 Months
  Mean change of hemoglobin A1c (in patients with Type 2 Diabetes (T2DM) from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cottam, MD, Principal Investigator — Bariatric Medicine Institute, Salt Lake City, UT; Walter Medlin, MD, Principal Investigator — Bariatric Medicine Institute, Salt Lake City, UT
Locations (1):
- Bariatric Medicine Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No